CLINICAL TRIAL: NCT06850558
Title: Patient's Satisfaction, Oral Health-related Quality of Life (OHRQoL) and Masticatory Efficiency of Mandibular Implant Supported Overdentures With Reduced Denture Base Extensions. A Within Subject Study
Brief Title: Patient's Satisfaction of Mandibular Implant Supported Overdentures With Reduced Denture Base Extensions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elgamal, Associate professor of prosthodontics, Mansoura University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A08011024RP
Record Dates: First submitted 2025-02-15; First posted 2025-02-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Patient Satisfaction Using Implant Retained Overdentures
Keywords: Mandibular implant overdentures y; Reduced denture base; Patient satisfaction; oral health-related quality of life; Masticatory efficiency
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: A within-subject study design was carried out; involving 20 completely edentulous participants aged 50-75 years, who received newly constructed conventional complete denture., implant overdenture (IOD) retained by bar attachment was constructed for each patient and were provided with two different overdenture designs: (1) firstly a fully extended denture base (FIOD) (2) then a reduced (partially extended) denture base (RIOD). Each patient allowed to wear each types of overdentures for a period of 3 months prior to evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fully extended denture base (Active Comparator): Patient allowed to wear fully extended overdenture base for a period of 3 months prior to evaluation after implants installation (four parallel implants) in the interforaminal region.
  Interventions: Procedure: Four parallel implants were installed in the interforaminal region
- partially extended denture base (Active Comparator): Patient allowed to wear partially (reduced) extended overdenture base for a period of 3 months prior to evaluation after implants installation (four parallel implants) in the interforaminal region.
  Interventions: Procedure: Four parallel implants were installed in the interforaminal region

INTERVENTIONS:
Procedure: Four parallel implants were installed in the interforaminal region — All participants administrated prophylactic antibiotics one day before implant placement and continued 7 days after surgery. Participants were asked to rinse their mouth with chlorhexidine mouthwash just before surgery and 7 days after surgery. Under local anesthesia, four implants were placed bilaterally in the interforaminal region. Four parallel implants (TioLogic, Dentaurum) were inserted in the inter-foraminal area using the submerged surgical approach and delayed loading protocol. By using the stereolithographic surgical guide the Implants were installed by the same surgeon with a minimum torque of 35 Ncm to give high initial stability. Relief was done in the mandibular denture over the implants and tissue conditioner (Visco-gel; DENTSPLY, Weybridge, UK) was used as a relining material. osseointegration was allowed to occur for a period of 3-6 months prior to final restoration.
  Other Names: Device (four titanium implant fixtures using submerged technique for implant installation protocol))

SUMMARY:
This study aimed to compare reduced (partially extended) denture bases with fully extended bases regarding patient satisfaction, oral health-related quality of life (OHRQoL), and masticatory efficiency.

A within-subject study design was carried out; involving 20 completely edentulous participants aged 50-75 years, who received newly constructed conventional complete denture. Four parallel implants were installed in the interforaminal region, implant overdenture (IOD) retained by bar attachment was constructed for each patient and were provided with two different overdenture designs: (1)firstly a fully extended denture base (FIOD) (2) then a reduced (partially extended) denture base (RIOD). Each patient allowed to wear each types of overdentures for a period of 3 months prior to evaluation. The following outcome measures were assessed: Patient satisfaction, the Oral Health Impact Profile (OHIP-14), and Chewing efficiency were assessed.

DETAILED DESCRIPTION:
Study Design This study is a within-subject comparison aimed at evaluating the effects of two different mandibular overdenture base designs: the Fully Extended Denture Base (FIOD) and the Reduced (Partially Extended) Denture Base (RIOD).

Study Protocol

1. Randomization: No randomization was done, the order of denture type presentation (was firstly fully extended then reduced design for each participant.
2. Adaptation Period: Participants were allowed a 3-months adaptation period for each Overdenture type to ensure familiarity and comfort.
3. Data Collection Schedule: Data for patient satisfaction, OHRQoL, and masticatory efficiency were collected at the end of each adaptation period. Data were collected at 3 months after use for each design, starting with FE design then RE.

Sample size and participants selection A total of 20 participants, aged 50-75 years, were recruited from the outpatient prosthodontic clinic, Faculty of Dentistry, Mansoura University. The sample size was determined based on a power analysis, aiming for an 80% power to detect significant differences at an alpha level of 0.05 and according to previous research in similar domains often utilized the same sample sizes.

Ethical Considerations The study was conducted in accordance with the Declaration of Helsinki, and ethical approval was obtained from the ethical committee, faculty of dentistry (A08011024RP). Informed consent was obtained from all participants prior to their involvement in the study. Participants were informed of their right to withdraw at any time without affecting their treatment.

Prosthetic and surgical procedures Newly constructed dentures with optimal flanges extension and balanced occlusal scheme using semi-anatomic acrylic teeth were delivered to all participants.

The participants were instructed to use the dentures for three months before implant placement to promote satisfactory neuromuscular control.

Following osseointegration duration, an open tray fixture level impression technique was performed using long transfer copings after splinting the copings with wire and auto polymerized resin (Duralay, Reliance Dental, Alsip, USA) to avoid movement during impression removal. The implant analogs were connected to the copings and the impression was poured. For Bar overdenture (BOD) prosthesis, plastic caps were screwed to bar abutments. Dolder bar joint plastic pattern (Dolder bar joint, Dentaurum) was lute to the caps with about 12mm distal cantilevers to reach the area of mandibular first molars. A 1-1.5 mm clearance space was kept between the ridge and the bar for cleaning reasons. The plastic bar was cast into cobalt-chromium and tried intraorally using Sheffield single screw test to check passivity. Titanium Dolder bar clips were fastened over the bar before processing of acrylic resin. The bar was then fitted with retentive clips or housings, which interfaced with the overdenture with fully extended base (FIOD), ensuring positive retention.

Following the 3 months period from FIOD mandibular implant overdenture use, data were collected then the overdenture was sent to the lab for reducing the denture base extension. The participant wore the mandibular implant overdenture with reduced denture base (Reduced Base Design) (RIOD) for another 3 months and the data were collected again .

Reduced (Partially Extended) Denture Base (RE): (R) A shorter base extending to the anterior portion of the mandible, designed to leave more space for tongue movement and enhance sensory feedback.

The design specifics are as follows:

- Geometric Configuration: The reduced base extends anteriorly to cover the anterior residual ridge while curving gently around the retromolar pad area. The posterior border is strategically positioned above the retromolar area to prevent impingement on the tissues and to allow for greater tongue space.

Dimensions: The dimensions of the reduced base were tailored individually based on each patient's anatomical features. The following measurements were taken into account:

* Anterior extension cut-off: 2 mm above the anterior alveolar ridge.
* Posterior limit: 5 mm anterior to the retromolar pad, which allows for optimal retention and avoids undue pressure on the underlying tissues.
* Buccal and lingual flanges were designed with a tapered profile to enhance aesthetic and functional features while maintaining adequate reinforcement.

Retention Mechanism: The overdenture was retained by four osseointegrated implants using bar-type attachments. These mechanisms were chosen for their ease of use and effective retention while allowing for minimal stress on the remaining alveolar ridge.

Statistical analysis:

Descriptive statistics were represented in the form of Mean ±Standard deviation (SD) .data was normally distributed as detected by Shapiro-wilk test. To compare patient satisfaction and OHRQoL scores between the 2 overdenture designs, Un-paired samples t-test was utilized as it was parametric data. While Wilcoxon signed-rank tests was applied to evaluate differences in masticatory efficiency measures as it was non-parametric data. The software package used for data analysis was SPSS® version 25 (SPSS Inc., Chicago, IL, USA). The level of significance was adjusted at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 75 years.
* Completely edentulous mandibular arch with adequate bone volume (≥10 mm in height and ≥ 6 mm in width at the implant site) and density to allow placement of 4 osseointegrated implants in the interforaminal region.
* Good general health, with no history of systemic diseases that would contraindicate implant placement or the use of overdentures.
* Presence of sufficient inter-arch space for overdenture construction and implant placement.
* No history of severe bruxism or parafunctional habits that could affect implant stability or prosthetic outcomes.
* Ability to understand and complete questionnaires regarding patient satisfaction and quality of life.
* Willingness to comply with the study protocol and attending follow-up visits.

Exclusion Criteria:

* History of temporomandibular joint disorders.
* Neurological disorders affecting masticatory function.
* Presence of uncontrolled systemic diseases.
* Cognitive impairments affecting the ability to provide informed consent.
* Severe bone resorption or contraindications for implant placement (e.g., insufficient ridge height or width).
* Presence of systemic diseases affecting oral health (e.g., uncontrolled diabetes, systemic inflammatory disorders).
* Inability to wear dentures for extended periods or intolerance to the study protocol

  7. Inability to wear dentures for extended periods or intolerance to the study protocol

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
I- Patient satisfaction | 3 months after each treatment
  Patient satisfaction was assessed using a questionnaire based on visual analog scale (VAS). Satisfaction was tested concerning comfort, esthetics, stability, speaking retention, general satisfaction. Patients were requested to mark their answer (amount of satisfaction) on a 100-mm line (with zero indicates not satisfied at all and 100 indicates to completely satisfied). Higher VAS scores showed high satisfaction and lower scores indicated low satisfaction. The mean of the answers (length of the lines from zero to the marks in mm) for every question was subjected to statistical analysis.
  All dimensions of this instrument were highly associated with the items of general satisfaction (Awad & Feine, 1998). The questionnaire was represented to the patients in Arabic
The oral health-related quality of life | 3 months after each treatment
  The oral health-related quality of life (OHRQoL) was assessed using the OHIP-14 oral health impact profile questionnaire, which consists of 7 categories: functional limitation, physical disability, physical pain

SECONDARY OUTCOMES:
Masticatory (chewing) efficiency | 3 months after each treatment
  The chewing efficiency was evaluated by a two-color mixing ability test following the technique illustrated by Schimmel et al utilizing Vivident Fruitswing chewing gum. Five gums samples prepared from two colored gums "Karpuz/Asai Üzümü" (gum3, Perfetti van Melle, Turkey): one with green color and the other with violet color were used in the chewing efficiency test. Patients were instructed to chew each sample (the violet side facing the palate) on their favored chewing side for 20 cycles. After chewing, the samples were prepared and labeled with random numbers . Both sides of the samples were scanned. The compound images were then evaluated with ViewGum software (dHAL Software, Greece). The software semiautomatically calibrate the hue value for each pixel after segmenting the image. Chewing efficiency was calculated using the variance of the hue (VOH) for each sample and the mean VOH for the 5 samples was subjected to statistical analysis. Good chewing efficiency produces more color

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Elgamal, PhD, Principal Investigator — Mansoura University; Abdallah M Ibrahim, PhD, Study Director — Mansoura University
Locations (1):
- Removable prosthodontics department,Faculty of dentistry,Mansoura university, #68 ElGomhoria Street, ElMansoura, Egypt., Al Mansurah, Eldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: No